CLINICAL TRIAL: NCT05714397
Title: Effectiveness of Cingal™ for Improving Pain Scores and Function in Anterior Knee Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Banff Sport Medicine Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB21-0205
Record Dates: First submitted 2023-01-17; First posted 2023-02-06 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cingal Injection (Experimental): Cingal will be administered by fellowship-trained physicians through ultrasound-guided injection using a 20-gauge needle into the joint space of the knee under sterile conditions. The needle track will be anesthetized with local anesthetic.
  Interventions: Device: Cingal

INTERVENTIONS:
Device: Cingal — A single Cingal injection will be administered by fellowship-trained physicians through ultrasound-guided injection using a 20-gauge needle into the joint space of the knee under sterile conditions. The needle track will be anesthetized with local anesthetic.

SUMMARY:
Anterior Knee Pain (AKP) is a common condition that can be challenging to treat effectively. The main goal of treatment regimens is to improve the function of the knee. However, treatment can be challenging due to the knee pain experience. Cingal™ contains hyaluronic acid (HA), which acts as a joint lubricant, and the corticosteroid triamcinolone hexacetonide (TH). Some studies have shown that Cingal™ can improve joint function and provide short-term pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 35 years
* Standard weight-bearing AP and skyline view knee x-rays
* Retropatellar or peripatellar knee pain for a minimum of 2 months
* Confirmed diagnosis of AKP that has failed to improve with a minimum of 6 weeks of conservative treatment (activity modification, supervised physiotherapy, exercise therapy, taping or bracing, NSAIDS)
* Pain aggravated by at least two of the following patellofemoral joint loading activities: squatting, running, ascending or descending stairs, or sitting with prolonged knee flexion.

Exclusion Criteria:

* X-ray evidence of knee osteoarthritis or fracture
* Meniscal or ligamentous injury assessed or suspected on clinical examination
* Previous knee surgery
* History of patellar instability
* Any contraindication to knee injection (overlying skin condition, joint infection, significant joint effusion, coagulopathy, previous adverse reaction, etc.)
* Known allergy to Cingal™ or its constituents
* Previous knee injection within the last 3 months
* BMI greater than 30 kg/m2
* Diabetes, inflammatory conditions (rheumatologic disease, ankylosing spondylitis), or concurrent medical conditions which may result in chronic pain or altered pain sensation
* Pregnant or breastfeeding
* Workers Compensation Board case
* Patient involved in litigation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
2D Kinematic Data | baseline, 6 weeks, 12 weeks
  Kinematic data will be collected at baseline and 6 and 12 weeks after administration of the Cingal™ injection. Outcome measures include ankle dorsiflexion at contact, maximum rear foot eversion, knee flexion at contact, knee adduction in late stance, and hip joint angle. In addition, the mean of three angle measurements for each parameter will be recorded.

SECONDARY OUTCOMES:
Strength Testing | baseline, 12 weeks
  A crane scale (strain gauge) will assess isometric strength testing of the quadriceps and hamstring muscles.
Biomechanical Assessment | baseline, 12 weeks
  The Drop Vertical Jump test will be used to assess dynamic valgus collapse of the knee.
Pain scores measured using a 100 mm Visual Analog Scale (VAS) | baseline, 4 days, 2 weeks, 4 weeks, 6 weeks, 12 weeks, 26 weeks
  The Pain VAS is anchored by 0, which corresponds to "no pain", and 10, which corresponds to the "worst possible pain".
Anterior knee pain using the Anterior Knee Pain Scale (AKPS) | baseline, 4 days, 2 weeks, 4 weeks, 6 weeks, 12 weeks, 26 weeks
  The AKPS is a 13-item knee-specific self-report questionnaire. It documents responses to six activities thought to be explicitly associated with anterior knee pain syndrome (walking, running, jumping, climbing stairs, squatting, and sitting for prolonged periods with knees bent), as well as symptoms such as limp, inability to weight bear through the affected limb, swelling, abnormal patellar movement, muscle atrophy and limitation of knee flexion. In addition, the AKPS asks about the duration of symptoms and the limb(s) affected. The maximum score is 100, and lower scores indicate greater pain/disability.
Symptoms of knee injury using the Knee Injury and Osteoarthritis Outcomes Score (KOOS) | baseline, 4 days, 2 weeks, 4 weeks, 6 weeks, 12 weeks, 26 weeks
  The KOOS is a knee-specific instrument developed to assess patients' opinions about their knee and associated problems.The KOOS assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
General activity rating using the Marx Activity Score | baseline, 4 days, 2 weeks, 4 weeks, 6 weeks, 12 weeks, 26 weeks
  The MARX Activity Rating Scale is a four-item activity rating scale where the patient is asked to rate how often they were able to perform each activity (e.g., running, cutting, decelerating, and pivoting) in their most healthy and active state. The four knee functions are rated on a 5-point scale of frequency (from 0 - 5) and scores are added up to a maximum of sixteen points, with a higher score indicating more frequent participation.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Hiemstra, MD PhD FRCSC, Principal Investigator — Banff Sport Medicine Foundation
Locations (1):
- Banff Sport Medicine, Canmore, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No